CLINICAL TRIAL: NCT04191694
Title: Chewing Gum for Prevention of Nausea and Vomiting After Elective Caesarean Section Under Spinal Anaesthesia: A Randomised Controlled Trial
Brief Title: Chewing Gum to Prevent Nausea and Vomiting After Caesarean Section Under Spinal Anaesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Petar Popivanov, Principal Investigator, Coombe Women and Infants University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-2019
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Chewing Gum; Ondansetron

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Patients will receive the standard dose of anti-emetic according to hospital practice (Ondansetron 4mg IV, intra-operatively)
  Interventions: Drug: Ondansetron 4 MG
- Chewing Gum (Active Comparator): Patients will receive the standard dose of anti-emetic according to hospital practice (Ondansetron 4mg IV, intra-operatively) they will also receive chewing in the recovery room and on the post-natal ward.
  Interventions: Other: Chewing Gum; Drug: Ondansetron 4 MG

INTERVENTIONS:
Other: Chewing Gum — Patients will be given a packet of chewing gum on arrival in the post-operative recovery room. They will be asked to start chewing gum in the recovery room and then asked to chew gum according to their preference over course of the following 24 hours.
  Arms: Chewing Gum
Drug: Ondansetron 4 MG — Ondansetron 4mg intravenously, intra-operatively as part of standard hospital caesarean section protocol

SUMMARY:
Our study aims to determine if there is a difference in a self-reported incidence of nausea and vomiting in women who are given chewing gum following elective caesarean section under spinal anaesthesia compared to those who do not receive chewing gum

DETAILED DESCRIPTION:
Caesarean section is one of the most commonly performed surgical procedures worldwide and the rate continues to rise. It is most often performed under regional anaesthesia, like spinal or epidural with long acting opioids such as spinal morphine added to improve postoperative pain in the first 24 hours.

However, nausea and vomiting is a common side effect of spinal morphine. Other risk factors for nausea and vomiting are patient related (female, non-smoker, history of post-operative nausea and vomiting [PONV] and/or motion sickness) and surgery related (spinal induced hypotension, blood loss, vagal stimulation, uterine exteriorisation, uterotonics, i.v. opioids etc). Risk assessment tools are available to estimate the risk of PONV for each patient.

The incidence of post-caesarean section nausea and vomiting at Coombe Women and Infants University Hospital is 28% and worldwide rates range from 21%-79%.

In the context of Enhanced Recovery After Surgery (ERAS), experiencing nausea and vomiting is distressing, reduces patient satisfaction by delaying early eating, drinking and mobilisation, interrupts bonding with the baby and prolongs hospital discharge.

It has been demonstrated that chewing gum is not inferior to 4 mg Ondansetron in treating nausea and vomiting post breast and laparoscopic surgery in female patients. It also has been shown to improve the return of gastrointestinal function after major surgery.

To our knowledge, no study has assessed the role of chewing gum for preventing nausea and vomiting after caesarean section under spinal anaesthetic.

Our study aims to assess whether or not chewing gum helps to reduce the self-reported incidence of nausea and vomiting in women undergoing caesarean section under spinal anaesthesia when compared to a control group who will not receive chewing gum.

There will be two arms of our study. Both arms will receive as standard Ondansetron 4mg intra-operatively.

One arm, the intervention arm, will then receive chewing gum, initially in the recovery room after their procedure and then will receive chewing gum to chew over the first 24 hours after their procedure according to their preference.

The second arm will not receive the chewing gum intervention.

Each arm will be followed up in the theatre recovery room after their procedure - determining any episodes of nausea or vomiting in the recovery room and the severity of episodes and whether any anti-emetic was given.

Each arm will also be followed up 24 hours later, asking them to report the number of episodes of nausea or vomiting they experienced in the 24 hours following their caesarean section and to assign the severity of their nausea or vomiting a number between 0-10,0 being none, 10 being most severe. The intervention arm will be asked how long they chewed chewing gum for in the first 24 hours after their procedure. The intervention arm will also be asked to rate their satisfaction with the intervention on a scale of 0-10, 0 being not satisfied, 10 being extremely satisfied.

All patients undergoing caesarean section will be considered for selection.

Patients will be identified at the pre-assessment clinic. At this review, patients will be identified for screening and will be assessed for eligibility.

The study will be discussed with them and they will be given a patient information leaflet.

Informed consent will be obtained prior to any study related procedures being undertaken.

The participants will be given a patient information leaflet prior to consent being taken. The information leaflet will be provided in simple and clear language. All patients will be informed of the objectives, benefits, risks and obligations imposed by the study. This discussion and consent will be performed in the pre-assessment clinic, thus allowing sufficient time to contemplate participation in the trial. Any questions or concerns will be addressed prior to consent being obtained. Informed consent will be obtained by an anaesthetic registrar on admission to hospital.

The study will be investigator led, single centre, randomised, unblind double arm comparator study

ELIGIBILITY:
Inclusion Criteria:

* Spinal Anaesthesia
* Elective
* Able and Agreeable to chew chewing gum in recovery room and in the first 24 hours
* Received Ondansetron 4mg IV intra-operatively

Exclusion Criteria:

* Type 1 Diabetes Mellitus
* Nausea and/or Vomiting on arrival to recovery room
* Post-partum haemorrhage >1000ml
* Ergometrine or Misoprostol intra-operatively
* Intravenous opioid intra-operatively

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the number of episodes of self-reported nausea | 24 hours post caesarean section
  Self-reported nausea described to investigator
The difference in the number of episodes of self-reported vomiting | 24 hours post caesarean section
  Self-reported number of episodes of vomiting described to investigator

SECONDARY OUTCOMES:
Episodes of nausea, vomiting or both in recovery room and at 24 hours after caesarean section. | 24 hours post caesarean section
  Number of episodes of nausea or vomiting experienced by women
Severity of nausea, reported as the worst episode in the last 24 hours | 24 hours post caesarean section
  Severity on a scale from 0-10, 0 being no nausea, 10 being extremely severe
Antiemetics in the first 24 hours after Caesarean section under spinal anaesthesia | 24 hours post caesarean section
  Number of doses of anti-emetic medication and the type of antiemetic given to women following their caesarean sections
Patient satisfaction with the intervention | 24 hours post caesarean section
  Patient satisfaction on 0 - 10 scale and Patient Reported Outcome Measure (PROM) - Obstetric Quality of Recovery (ObsQoR-11), currently part of the routine pain round

CONTACTS AND LOCATIONS:
Overall Officials: Terry Tan, Study Director — Coombe Women and Infants University Hospital
Locations (1):
- Coombe Women and Infants University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowe R, Irwin R, Browne G, Harbison M, Gallen S, Yore PJ, MacGearailt E, Popivanov P, Tan T. Chewing Gum for Prevention of Nausea and Vomiting After Elective Caesarean Section: a Pilot Randomised Controlled Trial. SN Compr Clin Med. 2022;4(1):257. doi: 10.1007/s42399-022-01332-9. Epub 2022 Nov 14. PMID 36404985